CLINICAL TRIAL: NCT07059585
Title: Does Perioperative Comprehensive Geriatric Assessment Reduce the Incidence of Postoperative Delirium in Older, Frail Patients Undergoing Elective Inpatient Surgery?
Brief Title: Preoperative Comprehensive Geriatric Assessment (CGA) and Postoperative Delirium
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Anesthesia Patient Safety Foundation (APSF) (Unknown)
Responsible Party: Principal Investigator, Elizabeth Mahanna Gabrielli, Associate Professor of Clinical Anesthesiology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230790
Record Dates: First submitted 2025-07-07; First posted 2025-07-11 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: CGA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CGA group (Experimental): Participants will receive the CGA intervention for up to 2 weeks
  Interventions: Behavioral: CGA
- Control Group (Other): Participants will receive standard of care treatment for up to 2 weeks
  Interventions: Other: control

INTERVENTIONS:
Behavioral: CGA — Participants will come once in person for the standard of care surgery. After the surgery, participants will receive delirium assessment questionnaires twice daily in the hospital for a duration of up to 7 days after surgery and, up to two sensory aids if required, one pair of eyeglasses as well as frequent orientation of physical and occupational therapy. On postoperative day 14, the subjects will be assessed for the same, whether at home or in-patient. The assessment completion could take up to an hour.
  Arms: CGA group
Other: control — Participants will come once in person for the standard of care surgery. After the surgery, participants will receive assessment questionnaires regarding perioperative delirium, twice daily in the hospital for a duration of up to 7 days after surgery. On postoperative day 14, the subjects will be assessed for the same, whether at home or in-patient. The assessment completion could take up to an hour.
  Arms: Control Group

SUMMARY:
The purpose of this research is to find out the best way to reduce delirium in frail, older patients undergoing planned surgery. Delirium is a state of confusion and difficulty concentrating that is temporary. Delirium may make the person anxious, angry, sleepy, not think clearly, or hallucinate. Being frail in medicine means that the body may not easily recover from a stressor, such as surgery. This study will determine if a detailed on-going evaluation by a Geriatrician, doctor who specializes in the care of older adults, after surgery is better at decreasing the risk of delirium than simply highlighting the patient's frailty in the electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Frailty as measured by the 5-modified frailty index (5-mFI) during the anesthesia preoperative assessment. The 5-mFI consists of 5 elements: 1-dependency for activities of daily living, 2-congestive heart failure within 30 days, 3-chronic obstructive pulmonary disease or pneumonia currently treated with antibiotics, 4-diabetes, and 5-hypertension. The diagnosis of frailty by the 5-mFI is based upon the presence of 2 or more of the elements.
2. Elective inpatient surgery with an expected LOS > 1 day;
3. Receiving general anesthesia
4. Adults who are unable to consent if they have a designated proxy able to consent

Exclusion Criteria:

1. Absence or withdrawal of informed consent,
2. Presence of current delirium
3. prisoners

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients of postoperative delirium (POD) as measured by confusion assessment measure (CAM) | up to 7 days
  The CAM score ranges from 1-4. Each score means the following:
  1. - acute onset or fluctuating course,
  2. - inattention,
  3. - altered mental status
  4. - disorganized thinking. The diagnosis of delirium by the CAM is based on the presence of features 1 and 2 and either 3 or 4.

SECONDARY OUTCOMES:
The proportion of patients who had a non-escalation of discharge level of care | 1 day (at the end of the intervention)
  The proportion of patients with non-escalation of discharge of level of care will be assessed by comparing the level of care of the location that the patient was living preoperatively to the level care to the location that the patient is discharged and will be considered present if the discharge level of care is the same or lower. Levels of care from highest to lowest are: long term acute care hospital > skilled nursing facility > rehabilitation center > assisted living > unassisted home living.
length of stay (LOS) | 1 day (at the end of the intervention)
  measured in number of days
prolonged length of stay (LOS) | 1 day (at the end of the intervention)
  measured in number of days
home delirium measured by CAM | up to 18 days
  measured by confusion assessment measure (CAM).Scores range from 1 through 4. Higher scores indicated higher confusion

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gabrielli, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No